CLINICAL TRIAL: NCT00434824
Title: A Multicenter, Randomized, Parallel-Group, Double-Blind, Placebo-Controlled Trial to Evaluate the Efficacy and Safety of Oral Administration of Different Doses of Org 538 in Symptomatic Aging Men With Androgen Deficiency
Brief Title: Effects of Andriol Testocaps in Symptomatic Late-Onset Hypogonadism (43203)
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 43203
Record Dates: First submitted 2007-02-12; First posted 2007-02-13 (Estimated); Last update posted 2015-04-16 (Estimated); Status verified 2015-04

CONDITIONS: Hypogonadism; Androgens
MeSH Terms: conditions — Hypogonadism | interventions — testosterone undecanoate

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Arm 1 (Active Comparator): Oral testosterone undecanoate (Andriol)
  Interventions: Drug: Oral testosterone undecanoate (Andriol)
- Arm 2 (Placebo Comparator): Placebo
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Oral testosterone undecanoate (Andriol) — treatment for 12 months with oral TU 80 mg/d, oral TU 160 mg/d or oral TU 240 mg/d in divided doses
  Other Names: Org 538
  Arms: Arm 1
Drug: Placebo — treatment for 12 months with placebo in divided doses
  Arms: Arm 2

SUMMARY:
In this study we have evaluated the effects of three different doses of oral testosterone undecanoate in aging men presenting with a combination of symptoms suggestive of hypogonadism and low blood levels of the male hormone testosterone.

Specifically, we have studied the effects on:

* symptoms suggestive of low testosterone levels
* blood testosterone and other hormone levels
* bone mass
* muscle mass and fat mass
* muscle strength
* prostate
* lipids, hematocrit

ELIGIBILITY:
Inclusion Criteria:

* Subjects were at least 50 years of age
* A body mass index (BMI) between 18 and 34 kg/m^2
* Symptoms of androgen deficiency (as indicated by a positive Androgen Deficiency in Aging Males (ADAM) questionnaire)
* Calculated free testosterone measurement of <0.26 nmol/L in the morning

Exclusion Criteria:

* History or current diagnosis of breast or prostate cancer
* any clinically significant abnormal finding on physical examination including the prostate
* Clinical symptoms of obstructive benign prostate hyperplasia (International Prostate Symptom Score (IPSS) >14)
* Prostate specific antigen (PSA) level > 4 ng/mL at screening
* Cause of androgen deficiency other than aging, e.g. 'classical' diagnosis of primary or secondary hypogonadism
* Hyperprolactinaemia or treatment with prolactin-lowering drugs
* History of known chronic polycythemia and/or hematocrit >50% at screening
* History or presence of severe sleep apnea
* Unstable or untreated endocrine disorders
* History or presence of clinically significant depression or other psychiatric disorder or any clinically relevant cardiovascular, cerebrovascular, endocrine, hepatic, renal or hematological disease, thromboembolism/thrombosis etc. which, in the opinion of the investigator, might compromise the subject's participation in the trial
* Use of medication that would interfere with the efficacy and safety objectives of the trial

Min Age: 50 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 322 (Actual)
Dates: Start 2001-11; Primary Completion 2004-07 (Actual); Study Completion 2004-07 (Actual)

PRIMARY OUTCOMES:
Change from baseline on the total score of the AMS rating scale | Month 6

SECONDARY OUTCOMES:
Effects on AMS rating scale, bone mineral density, bone markers, muscle and fat mass, muscle strength, hematocrit, endocrine parameters, PSA, IPSS and lipids | Month 12

REFERENCES:
- [Derived] Meuleman EJ, Legros JJ, Bouloux PM, Johnson-Levonas AO, Kaspers MJ, Elbers JM, Geurts TB, Meehan AG; Study 43203 Investigators. Effects of long-term oral testosterone undecanoate therapy on urinary symptoms: data from a 1-year, placebo-controlled, dose-ranging trial in aging men with symptomatic hypogonadism. Aging Male. 2015;18(3):157-63. doi: 10.3109/13685538.2015.1032925. Epub 2015 Jun 1. PMID 26030346
- [Derived] Bouloux PM, Legros JJ, Elbers JM, Geurts TB, Kaspers MJ, Meehan AG, Meuleman EJ; Study 43203 Investigators. Effects of oral testosterone undecanoate therapy on bone mineral density and body composition in 322 aging men with symptomatic testosterone deficiency: a 1-year, randomized, placebo-controlled, dose-ranging study. Aging Male. 2013 Jun;16(2):38-47. doi: 10.3109/13685538.2013.773420. Epub 2013 Apr 12. PMID 23581697